CLINICAL TRIAL: NCT02177929
Title: Study About Acting of Adaptive Sport in Musculoskeletal, Cardiovascular System and the Quality of Life of Individuals With Spinal Cord Injury Through Biomedical Instrumentation
Acronym: Adaptive sport
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universidade do Vale do Paraíba (Other)
Responsible Party: Principal Investigator, Izabela dos Santos Mendes, Study about acting of adaptive sport in musculoskeletal, cardiovascular system and the quality of life of individuals with spinal cord injury through biomedical instrumentation, Universidade do Vale do Paraíba
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CAAE: 18353613.0.0000.5503
Record Dates: First submitted 2014-06-18; First posted 2014-06-30 (Estimated); Last update posted 2014-06-30 (Estimated); Status verified 2014-06

CONDITIONS: Adaptive Sport in Spinal Cord Injury
Keywords: Spinal cord injury,; adaptive sport,; dynamometry,; electromyography,; force platform.
MeSH Terms: conditions — Spinal Cord Injuries

ARMS (1):
- adapted canoeing, handbike, conventional physiotherapy (Experimental): Individuals are divided into three groups: one group adapted canoeing, one group of handbike and one grup of conventional physiotherapy.
  Interventions: Other: adapted canoeing, hadbike and conventional physiotherapy

INTERVENTIONS:
Other: adapted canoeing, hadbike and conventional physiotherapy — The subjects adapted canoeing group will practice on the kayak and rowing exercises associating with ball.
  The individuals in the group will handbike workouts outdoors and surpassing cirucuitos mounted with cones.
  Individuals in the conventional physiotherapy group will make stretching and strengthening exercises.

SUMMARY:
The hypothesis is to the fulfillment of canoeing, handbike and conventional physiotherapy activities the groups could show improvement in muscle strength of the arms, decreased resistance of the lower limbs (spasticity), improved trunk balance and movements of the upper limbs, improves cardiovascular function, bone health, and consequently improve the quality of life.

ELIGIBILITY:
Inclusion Criteria:

* aged 15-40 years
* of both sexes
* with injury time over 8 months, who present spasticity in the lower limbs up to grade 2 according to the scale of Ashwoth modified patient with paraplegia or paraparesis in thoracolumbar level (lower than T2) levels.

Exclusion Criteria:

* age over 40 years
* lesion less than 8 months
* above T2 lesions
* musculoskeletal disorders such as deformity
* severe contracture
* previously diagnosed cardiovascular abnormalities or risk factors such as hypertension
* diabetes and obesity, use of medications and cardiopressant cardioestimuladoras, smoking and alcoholics.
* For individuals who participate in the group canoeing and by adapting the pool will still include the following exclusion criteria:

  * decubitus ulcers
  * fungal infections
  * urinary incontinence
  * inflammatory processes and neoplasms.

Ages: 15 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 45 (Estimated)
Dates: Start 2013-04; Primary Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Evaluate of torque | Data collection for 11 months.
  The isokinetic dynamometer Biodex System will be used to evaluate the torque of biceps and triceps brachii of the dominant limb. The protocol will be conducted in 5 replicates in concentric isokinetic mode for flexion and extension of the elbow. The range of motion is from 80 to elbow extension, adopting as the 0 ° position in which the longitudinal center line of the lever arm of the dynamometer will remain parallel to the ground. The forearm of individuals remain in neutral pronation-supination, the shoulder joint is maintained at 45 ° of flexion and abduction. The unit of measure will be N.m
Evaluation of resistance to stretching of the flexors and extensors knee | For 11 months
  Individuals will be submitted to test resistance to stretching of the flexors and extensors knee of the dominant leg, through isokinetic dynamometer Biodex System. To perform the test the individual remain seated and stabilized in equipment with hip and knee flexed to 90°. The lever arm is positioned at 2 cm from the malleoli (medial and lateral) axes of the ankle and the dynamometer coincide with the axis of movement of flexion-extension of the knee. After positioning, the dynamometer in passive mode will be triggered to perform 5 repetitions of knee flexion-extension in an angular velocity of 120 °/s, and range of motion of 90°. Individuals will be instructed not to perform any kind of contraction or voluntary movement. The unit of measure is N.m.
Electromyography of knee extensors | 11 months
  Simultaneously, the evaluation of the tone of the lower limbs through dynamometry muscle activity will be captured by means of EMG. Electromyographic variables are captured in relation to the quadriceps muscle group of the dominant limb. Surface electrodes are placed on the muscle belly of the rectus femoris, vastus medialis and vastus lateralis according to the recommendations of SENIAM (Surface Electro MyoGraphy for the Non-Invasive Assessment of Muscles). The EMG signal is acquired with a sampling frequency of 2000 Hz and unit reader of channels in microvolts. The data are normalized by the average of electromyographic signals during passive movement performed by isokinetic dynamometer.
Electromyography of erector trunk | 11 months
  Electromyographic variables are also captured in relation to the erector muscles of the trunk. Surface electrodes are placed on the muscle belly (bilaterally), 2 cm from the vertebra, corresponding to one segment above the level of the lesion for each group analyzed point. The EMG signal is acquired with a sampling frequency of 2000 Hz and unit reader of channels in microvolts. The data are normalized by the average of electromyographic signals obtained during the stabilization of the trunk through the force platform test, described below.
Evaluation of trunk balance | 11 months
  Simultaneously, the EMG of the erector muscles of the trunk, the trunk balance will be assessed using a force platform, EMG system brand in Brazil, which has four load cells and acquisition frequency of 2000 Hz This platform analyzes anteroposterior oscillation. In the evaluation, patients remain in sitting under the platform with outstanding lower limbs and upper limbs along the body for 30 seconds with eyes open and then with eyes closed position. The unit of measure will be Kgf.
kinematic analysis | 11 months
  To analyze the movements of the upper limbs markers will be fixed in the following anatomical landmarks: lateral center of the shoulder joint, lateral trunk, elbow, wrist and fifth metacarpal head of the dominant limb. The regions where the markers will be fixed previously cleaned with cotton and alcohol to remove the natural oils from the skin, allowing for better fixation of the markers. The videos will be played during activities of canoeing and handbike so adapted to the collection. The video camera will be positioned laterally to the individual. For canoeing gathering will be held at the clinic hydrotherapy and movement of boating pool is played similarly for 2 min, with guy in kayak. And for analyzing the movements performed for handbike, subjects will be shot while performing movements with handbike on a roll for 2 minutes. The joint angles of the shoulder, elbow and wrist, and the pace of movement will be analyzed.
Analysis of heart rate varibilidade | 11 months
  Data will be collected through the heart monitor Polar RS 800 then will be transferred to a microcomputer equipped with Polar ProTrainer software. The signal will be filtered and exported to Matlab 6.1 to perform the Continuous Wavelet Transform (TWC) in order to obtain for the spectral analysis variables: low frequency - LF = Low Frequency, 0.04-0.15 Hz and high frequency - HF = High Frequence, 0.15-0.4 Hz; and a temporal analysis variables: HR, RR, SDNN, RMSSD and PNN50.
Evaluation of quality of life | 11 months
  To assess the quality of life questionnaire World Health Organization Quality of Life in its shortened version - WHQOL-BREF is used. This instrument consists of 26 questions, of which 24 are divided into four domains: physical, psychological, social relationships and environment, in addition to these four areas, the instrument features two general questions: one refers to the perception of quality of life and other satisfaction with health. All responses are composed of graduated scale with scores ranging from one to five points.

SECONDARY OUTCOMES:
Data Analysis | 6 months
  For data analysis, dynamometry and electromyography (EMG) is used to EMGworks Program 3.1.1.1 Analysis of Delsys.
  To dynamometry, delete the first and last repetition and will be calculated for the mean peak torque of upper limb and root mean square (RMS - English root mean square) for resistance to passive movement of the lower limb. For electromyographic analysis, will be using a 4th order bandpass filter (20-400 Hz) and the RMS value is calculated for each signal.
  The heart rate variability will be analyzed by Wavelet raw state.
  For data analysis of quality of life an application Excel is used.
  For the remaining data will be given on how best analysis.
  The statistical analysis will be performed using the program Bioestat

CONTACTS AND LOCATIONS:
Locations (1):
- Universidade do Vale do Paraíba, São José dos Campos, São Paulo, Brazil